CLINICAL TRIAL: NCT00002754
Title: PHASE I STUDY OF MONOCLONAL ANTIBODY FRAGMENT 131I MEL-14 F(AB')2 VIA SURGICALLY CREATED CYSTIC RESECTION CAVITY IN THE TREATMENT OF PATIENTS WITH PRIMARY OR METASTATIC MALIGNANT MELANOMA AND OTHER BRAIN TUMORS
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Primary or Metastatic Melanoma or Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000064690; DUMC-0334-99-2R6; DUMC-219-96-2R3; DUMC-302-97-2R4; DUMC-308-98-2R5; NCI-V96-1071
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors; Melanoma (Skin); Metastatic Cancer
Keywords: recurrent adult brain tumor; adult glioblastoma; stage IV melanoma; tumors metastatic to brain; childhood high-grade cerebral astrocytoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; recurrent childhood cerebral astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Melanoma; Neoplasm Metastasis; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma

INTERVENTIONS:
Biological: monoclonal antibody Me1-14 F(ab')2

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to determine the effectiveness of monoclonal antibody therapy in treating patients who have primary or metastatic melanoma or brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and maximum tolerated dose of iodine-131-labeled monoclonal antibody fragment ME1-14 F(ab')2 administered intracystically in patients with recurrent or newly diagnosed primary or metastatic malignant melanoma or other brain tumors. II. Identify any objective therapeutic responses to this treatment.

OUTLINE: All patients receive a fixed dose of monoclonal antibody fragment ME1-14 F(ab')2 via an intralesional catheter; cohorts of 3-6 patients receive escalating doses of isotope conjugated to the antibody until the maximum tolerated dose is determined. Patients with newly diagnosed disease at entry may receive additional therapy with external-beam radiotherapy beginning 4 months after radioimmunotherapy (or sooner if disease progression occurs). Patients with recurrent disease at entry are followed without further therapy for at least 4 months after radioimmunotherapy; alternative therapy may be offered upon progression. All patients are followed at 4, 8, 16, and 24 weeks after treatment, then every 12 weeks for 1 year.

PROJECTED ACCRUAL: Three to six patients will be entered at each dose studied.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary or metastatic malignant melanoma OR Histologically confirmed supratentorial malignant brain tumor Newly diagnosed or recurrent primary or metastatic tumor Eligible primary histologies, including but not limited to: Glioblastoma multiforme Mixed anaplastic glioma Anaplastic astrocytoma Other astrocytoma Gliosarcoma Anaplastic oligodendroglioma The following excluded: Diffusely infiltrating tumors Multifocal tumors Infratentorial tumors Subependymal spread No measurable enhancing lesion extending more than 1 cm beyond margins of surgical cavity on contrast-enhanced CT or MRI performed within 72 hours after resection Intralesional catheter placed at resection Patency of catheter demonstrated by radiolabeled albumin flow Reactivity of neoplastic cells with intact Me1-14 IgG2a or Me1-14 F(ab')2 demonstrated by immunohistology with polyclonal rabbit antibody or monoclonal mouse antibody

PATIENT CHARACTERISTICS: Age: 3 and over Performance status: Karnofsky 50%-100% Hematopoietic: Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST less than 1.5 times normal Alkaline phosphatase less than 1.5 times normal Renal: Creatinine less than 1.2 mg/dL Other: Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 weeks since antineoplastic chemotherapy unless unequivocal tumor progression Endocrine therapy: Concurrent corticosteroids allowed at lowest possible dose and stable for at least 10 days prior to entry Radiotherapy: At least 3 months since radiotherapy to site of measurable disease within the nervous system unless unequivocal tumor progression Surgery: See Disease Characteristics

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 1993-02; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell D. Bigner, MD, PhD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States